CLINICAL TRIAL: NCT05507086
Title: Blue Sweat - Infectious Pseudochromdrosis Caused by Bacillus Cereus
Brief Title: Infectious Pseudochromdrosis Caused by Bacillus Cereus
Acronym: Blue sweat
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Christoffer Aam Ingvaldsen, Researcher, University Hospital, Akershus
Other Study IDs: IPCH2
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Infectious Disease; Bacterial Overgrowth; Pigment Deposition
Keywords: Infectious pseudochromhidrosis; Chromhidrosis; Sweat; Bacillus cereus
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Skin swabs for microbiological examinations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Antimicrobial therapy — Antimicrobial therapy

SUMMARY:
Twelve patients with blue sweat (infectious pseudochromhidrosis) caused by Bacillus cereus.

DETAILED DESCRIPTION:
Case series/observational study. Twelve patients with blue sweat (infectious pseudochromhidrosis) caused by Bacillus cereus. Demography, clinical presentation, diagnosis, treatments, microbiology and causality.

ELIGIBILITY:
Inclusion Criteria:

* Infectious pseudochromhidrosis caused by Bacillus cereus

Exclusion Criteria:

* Other types of blue chromhidrosis

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Twelve patients with blue sweat (infectious pseudochromhidrosis) caused by Bacillus cereus
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Remission | 1 year
  Descriptive / physical examination
Repeated bacteriological swab | 1 year
  Repeated bacteriological swab if uncertainty in terms of complete remission

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Microbiology, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No